CLINICAL TRIAL: NCT05495295
Title: An Adaptive First-in-human Trial of PhOx430, a First-in-class Acetylglucosaminyltransferase V Inhibitor, in Patients With Advanced Solid Tumours (PhAST Trial)
Brief Title: First-in-human Trial of PhOx430, a First-in-class Acetylglucosaminyltransferase V Inhibitor, in Advanced Solid Tumours
Acronym: PhAST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Phost'In Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHOX-CLI_001; 2021-004170-55 (EudraCT Number)
Record Dates: First submitted 2022-07-27; First posted 2022-08-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Malignant Tumor; Advanced Solid Tumor; Glioblastoma Multiforme; Metastatic Cancer
MeSH Terms: conditions — Neoplasms; Glioblastoma; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: First-in-human clinical trial, including two parts: a dose escalation phase (part I) which will enroll patients with non-selected tumour types, followed by a cohort expansion phase (part II) in selected tumour types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced Solid Tumours (Experimental): First-in-human clinical trial of the acetylglucosaminyltransferase V inhibitor PhOx430 in patients with advanced solid tumours. The trial includes two parts, a dose escalation phase (part I) which will enroll patients with non-selected tumour types, followed by a cohort expansion phase (part II) in selected tumour types:
  * Glioblastoma Multiforme (GBM)
  * Triple Negative Breast Cancer (TNBC)
  * Selected solid tumours
  Interventions: Drug: PhOx430

INTERVENTIONS:
Drug: PhOx430 — A standard 3 + 3 design will be followed. PhOx430 will be administered orally twice a day (bid), at a 12-hour interval, continuously in cycles of 21 days. At each dose level (DL), three patients will be included and the first patient will be observed for at least 21 days before enrolling the following two. Three additional patients will be enrolled at each DL if a DLT is observed in the first three patients.
  A maximum of 4 increasing Dose Levels are foreseen (10, 20, 40 and 70 mg/kg/day), and PhOx430 will be administered in two doses at a 12-hour interval.
  Other Names: Dose Escalation Phase - STEP 1 and STEP 2
Drug: PhOx430 — The implementation of this cohort (Step 3) was decided by the Protocol Steering Committee (PSC) based on clinical and pharmacokinetic data obtained in Steps 1 and 2. Six patients will be enrolled, who will receive PhOx430 orally thrice a day (tid) at a -6-hour interval over 12 hours for 21 days, and then, starting from day 22, four times a day (qid) at a 4-hour interval over 12 hours, continuously in cycles of 21 days. PhOx430 will be taken in single doses of 1,200 mg to patients weighing ≥ 50 kg and of 600 mg to patients weighing < 50 kg, with no requirement for a full or empty stomach. The first patient will be observed after treatment start for at least 21 days before enrolling the following two. After the third patient is observed for 21 days after treatment start, 3 additional patients will be enrolled without waiting time between them. If the daily dose tested with the tid schedule is not deemed safe, the flat dose will be tested twice a day (bid) at a 12-hour interval.
  Other Names: Dose Escalation Phase - STEP 3 (Dosing-optimization Cohort)

SUMMARY:
The PhAST Trial is an adaptive first-in-human clinical trial of the acetylglucosaminyltransferase V inhibitor PhOx430 in patients with advanced solid tumours conceived and designed with the contribution of the Gianni Bonadonna Foundation, a non-profit academic research institution aimed at promoting therapeutic innovation in oncology.. The trial includes two parts, a dose escalation phase which will enroll patients with non-selected tumour types, followed by a cohort expansion phase in selected tumour types.

DETAILED DESCRIPTION:
The PhAST Trial is a first-in-human clinical trial of the acetylglucosaminyltransferase V inhibitor PhOx430 in patients with advanced solid tumours. The trial includes two parts, a dose escalation phase (part I) which will enroll patients with non-selected tumour types, followed by a cohort expansion phase (part II) in selected tumour types.

POPULATION:

Adult patients with advanced or metastatic solid malignancies with radiologically documented progression on a previous line of treatment and for which effective treatment options do not exist.

DOSE ESCALATION'S PRIMARY OBJECTIVE:

To determine the Maximal Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) of PhOx430 in patients with advanced solid tumours

DOSE ESCALATION'S SECONDARY OBJECTIVE:

1. to determine the safety and tolerability profile of PhOx430 at increasing dose levels;
2. to characterize the pharmacokinetic (PK) profile of PhOx430, including food effect on drug disposition;
3. to evaluate the antitumour activity of PhOx430.

   DOSE ESCALATION'S EXPLORATORY OBJECTIVE:
4. to characterize the pharmacodynamics (PD) effect of PhOx430 on blood, urine and tumour samples collected before and after treatment;
5. to identify predictive response biomarkers by profiling responsive patterns.

DOSE EXPANSIONS' PRIMARY OBJECTIVE:

To better characterize the safety and tolerability profile of PhOx430 given at the RP2D in three cohorts of patients affected by 1) glioblastoma multiforme (GBM), 2) triple-negative breast cancer, and 3) selected types of solid tumours.

DOSE EXPANSION'S SECONDARY OBJECTIVE:

1. to characterize the pharmacokinetic (PK) profile of PhOx430 at the RP2D.
2. to evaluate the antitumour activity of PhOx430 in the specific tumour types selected for the dose expansion cohorts.

   DOSE EXPANSIONS' EXPLORATORY OBJECTIVE:
3. to characterize the pharmacodynamic (PD) effect of PhOx430 on blood, urine and tumour samples collected before and after treatment;
4. to identify predictive response biomarkers by profiling responsive patterns.

STUDY DESIGN AND TREATMENT PLAN:

Dose Escalation Phase - STEP 1-2: a standard 3 + 3 design will be followed. PhOx430 will be administered orally twice a day (bid), at a 12-hour interval, continuously in cycles of 21 days. At each dose level (DL), at least three patients will be included and the first patient will be observed for at least 21 days before enrolling the following two.

Dose Escalation Phase - STEP 3 (Dosing-optimization Cohort): The implementation of this Dosing-optimization cohort (Step 3) was decided by the Protocol Steering Committee (PSC) based on clinical and pharmacokinetic data obtained in Steps 1 and 2. Six patients will be enrolled, who will be administered a flat dose of PhOx430 (1,200 mg by patients weighing ≥ 50 kg and of 600 mg by patients weighing < 50 kg) orally thrice a day (tid) for 21 days, and then, starting from day 22, four times a day (qid), continuously in cycles of 21 days. The first patient will be observed after treatment start for at least 21 days before enrolling the following two. After the third patient is observed for 21 days after treatment start, three additional patients will be enrolled without waiting time between them. In case the daily dose tested with the tid schedule is not deemed safe, the flat dose of PhOx430 will be tested twice a day (bid).

Cohort Expansion Phase: in the cohort expansion phase, the safety profile of PhOx430 will be further characterized by testing the RP2D in three parallel cohorts of patients affected by glioblastoma multiforme (GBM) (cohort 1), triple-negative breast cancer (TNBC) (cohort 2), and solid tumour types selected by the Protocol Steering Committee (PSC) on the basis of preclinical pharmacological data and of the antitumour activity observed during the Dose Escalation Phase if any (cohort 3), respectively. Cycles will be of 21 days.

ESTIMATED TRIAL DURATION and SAMPLE SIZE:

Dose Escalation Phase Step 1,2,3: approximately 1.5 years Expansion Phase: approximately 1.5 years. The end of trial is defined as 30 days after the last dose of the last enrolled patient.

The following numbers of patients are foreseen: up to 149 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of cancer.

   1. Dose escalation phase: patients with any solid tumour type or histology.
   2. Expansion cohort 1: Patients affected by GBM.
   3. Expansion cohort 2: Patients with triple-negative breast cancer (TNBC), defined as estrogen receptor (ER) negative (< 1% of nuclei reacting for ER in IHC), progesterone receptor (PgR) negative (< 1% of nuclei reacting for PgR in IHC), HER2 negative (IHC score = 0 or 1 or ICH score = 2 with FISH negative for HER2 overexpression. If only FISH was performed, negative result for HER2 overexpression).
   4. Expansion cohort 3: Patients affected by solid tumour types selected by the PSC, on the basis of preclinical pharmacological data and of the antitumour activity observed during the dose escalation phase if any.
2. Radiologically documented progressive disease after at least one prior treatment for metastatic/advanced disease.
3. Lack of standard effective treatment options.
4. Female or male patients of ≥ 18 years and ≤ 80 years
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1. For GBM patients: Karnofsky Performance Status ≥ 50%.
6. Recovery from acute reversible toxicities of previous treatment to Grade ≤ 1.
7. Tumour tissue accessible for repeated biopsies (except GBM patients).
8. For GBM patients: stable dose of corticosteroids for > 5 days before the baseline MRI scan.
9. For non-GBM patients: Measurable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST) guideline V1.1 (specifically, no ascites, pleural or pericardial effusions, osteoblastic bone metastases, or carcinomatous lymphangitis of the lung as the only lesion). For GBM patients: Measurable disease as defined by RANO criteria.
10. Adequate bone marrow function defined as:

    1. absolute neutrophil count ≥ 1.5 x 109/L (being > 2 weeks off hematopoietic growth factors),
    2. platelet count ≥ 100 x 109/L,
    3. hemoglobin ≥ 9 g/dl without transfusions in the last 2 weeks.
11. Adequate hepatic function defined as:

    1. total bilirubin < 1.5 x the upper limit of normal (ULN),
    2. ALT /AST (SGPT/SGOT) < 3 x ULN (< 5 x ULN in the presence of known hepatic metastases),
12. Adequate renal function defined as estimated glomerular filtration rate (eGFR) of > 50 ml/min/1.73 m2 according to the CKD-EPI formula.
13. Adequate coagulation, defined as INR < 1.5 and aPTT < 1.5 × ULN. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
14. Written informed consent obtained prior to any trial-specific screening procedures.
15. Life expectancy of at least 3 months
16. Women of childbearing potential must have a negative serum pregnancy test obtained within 28 days prior to treatment start; in addition, the negative result is to be confirmed by a repeat urine or serum pregnancy test within 72 hours before study treatment start if the screening test was performed earlier.
17. Female patients who are not postmenopausal ("postmenopausal" defined as ≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus) must agree to practice a highly effective method of contraception throughout the study for at least 6 months after the last dose of study drug. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl Index of < 1% per year when used consistently and correctly. Sexual abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
18. Male patients must agree to remain sexually abstinent or use a condom during the treatment period and for at least 90 days after the last dose of study drug.
19. Patients must be able to take IMP at home and to properly use the provided dosing device.

Exclusion Criteria:

1. Major surgery, chemotherapy, radical radiotherapy, investigational agents, or other anticancer therapy in the last 4 weeks before treatment start.
2. For all patients with the exception of GBM patients: active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (subjects with a history of CNS metastases or cord compression are allowable if they have been definitively treated and have been clinically stable for at least 3 months, and off steroids or anticonvulsants, before day 1 treatment).
3. For GBM patients: disease progression within three months following last prior radiation therapy.
4. Inability or unwillingness to swallow.
5. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the IMP (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome)
6. Any other cancer within 3 years prior to enrolment, with the exception of adequately treated carcinoma in situ of the cervix uteri, or adequately treated basal or squamous cell carcinoma of the skin.
7. Significant liver disease, including active viral, alcoholic or other hepatitis and cirrhosis.
8. History of HIV infection, active hepatitis B (chronic or acute), or hepatitis C infection. Patients with past or resolved hepatitis B infection (defined as having a negative HBsAg test and positivity for antibodies for hepatitis B core antigen [anti-HBc]) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA
9. Severe infections within 4 weeks prior to enrolment.
10. Patients with a history of central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and precluding informed consent or adversely affecting compliance with study drug.
11. Baseline left ventricular ejection fraction (LVEF) < 50% by echocardiography or multi-gated scintigraphic scan (MUGA)
12. Other current severe, uncontrolled systemic disease
13. Treatment with CYP3A4/5 inhibitors within 5 drug elimination half-lives before study treatment start and/or inability or unwillingness to avoid such medications during study treatment
14. Known hypersensitivity to any study drug components
15. Pregnant or lactating women
16. Patients deprived from liberty (for patients enrolled in France only)
17. Patients who are not affiliated to a social security scheme or are not beneficiaries of such a scheme (for patients enrolled in France only)
18. Adults under legal protection or unable to give their informed consent (for patients enrolled in France only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
DOSE ESCALATION PRIMARY OUTCOME (Dose Limiting Toxicities (DLTs)) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  Dose Limiting Toxicities (DLTs)
DOSE EXPANSION PRIMARY OUTCOME (treatment-emergent Adverse Events) | Through study completion, up to 5 years
  Incidence, severity and seriousness of treatment-emergent Adverse Events (AEs)

SECONDARY OUTCOMES:
DOSE ESCALATION SECONDARY OUTCOME #1 (treatment-emergent Adverse Events) | Through study completion, up to 5 years
  Incidence, severity and seriousness of treatment-emergent Adverse Events (AEs)
DOSE ESCALATION SECONDARY OUTCOME #2 (Plasma concentration levels of PhOx430) | During Cycle1 and Cycle 2 (each cycle is 21 days)
  Plasma concentration levels of PhOx430
DOSE ESCALATION SECONDARY OUTCOME #3 (Objective response rate) | Through dose escalation completion, an average of 1 year
  Objective response rate (ORR)
DOSE EXPANSION SECONDARY OUTCOME #1 (Plasma concentration levels of PhOx430 ) | During Cycle1 and Cycle 2 (each cycle is 21 days)
  Plasma concentration levels of PhOx430
DOSE EXPANSION SECONDARY OUTCOME #2 (Objective response rate) | Through dose expansion completion, an average of 1.5 year
  Objective response rate (ORR)
DOSE ESCALATION SECONDARY OUTCOME #4 (progression-free survival) | Through study completion, up to 5 years
  progression-free survival (PFS)
DOSE ESCALATION SECONDARY OUTCOME #5 (overall survival) | Through study completion, up to 5 years
  overall survival (OS)
DOSE EXPANSION SECONDARY OUTCOME #3 (progression-free survival) | Through study completion, up to 5 years
  progression-free survival (PFS)
DOSE EXPANSION SECONDARY OUTCOME #4 ( overall survival) | Through study completion, up to 5 years
  overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Herrera, MD, Study Director — Phost'In Therapeutics; Diego Tosi, MD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (4):
- Institut du Cancer de Montpellier, Montpellier, France
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Unità Sanitaria Locale - IRCCS di Reggio Emilia, Reggio Emilia